CLINICAL TRIAL: NCT00647023
Title: Incretin Secretion in Women With Polycystic Ovary Syndrome (PCOS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Incretin secretion in women with PCOS, Pernille Fog Svendsen
Purpose: Basic Science
Other Study IDs: Incretins and PCOS
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: metformin — 1000 mg metformin x 2 daily during 8 months

SUMMARY:
The incretin hormones are secreted from the gastrointestinal tract in response to nutrient ingestion, and are responsible for 70 % of insulin secretion in response to glucose. The incretin response is attenuated in subjects with type 2 diabetes and other conditions associated with insulin resistance. Polycystic ovary syndrome (PCOS) is characterised by irregular periods and increased androgen levels. It is the most common endocrine disorder amongst young women at fertile age, and the most common cause of female infertility. Insulin resistance plays an important role in the development of the disease, and women with PCOS are at increased risk of developing tyoe 2 diabetes. the incretin hormones have not previously been investigated in women with PCOS, and the purpose of the present study was to investigate the secretion of the two most important incretin hormones Glucose-like peptide-1 (GLP-1) and Glucose dependent insulinotropic peptide (GIP) during a three hour oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who fulfill the Rotterdam criteria for PCOS. Age 18-38

Exclusion Criteria:

* Other endocrine diseases or diseases known to influence glucose/insulin/fat metabolism
* Oral contraceptive administration within three months of study start

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2004-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)